CLINICAL TRIAL: NCT06333847
Title: Are Multimorbidity and Related Factors Associated With Non-response Bias in Patients With Spinal Pain? - A Prospective Cohort Study
Brief Title: Are Multimorbidity and Related Factors Associated With Non-response Bias in Patients With Spinal Pain?
Status: Active, not recruiting | Type: Observational
Sponsor: Jacob Christiansen Gandløse (Other)
Responsible Party: Sponsor-Investigator, Jacob Christiansen Gandløse, Principal investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: K2023-059
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Back Pain; Low Back Pain; Neck Pain; Comorbidities and Coexisting Conditions
Keywords: back pain; low back pain; Neck pain; Comorbidities; coexisting conditions; Multimorbidity; Non-response bias; Successive wave-analysis
MeSH Terms: conditions — Back Pain; Low Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: Patients who responded to the first invitation to participate
- Group 2: Patients who responded to the second invitation to participate
- Group 3: Patients who responded to the third invitation to participate
- Group 4: Patients who did not respond to inviations to participate
- Group 5: Patients who responded to invitations to participate and thus an amalgamation of the people from groups 1, 2 and 3

SUMMARY:
The study aims to explore if non-response bias exists among individuals with chronic back pain, focusing on the impact of chronic disease count, treatment burden from multimorbidity, and health-related quality of life. Data is gathered from patients at Aalborg University Hospital's Rheumatology Department via electronic means and medical records. The analysis comprises two-wave assessments, investigating disparities among patients responding to study invitations based on response patterns: first, second, or third invitation responses. Utilizing baseline data, a one-way ANOVA is employed to detect potential between-group variations in the mentioned factors. Subsequently, a repeated measures ANOVA is conducted to evaluate differences among groups over time. Additionally, statistical analyses are conducted to scrutinize variances in age and gender distribution between respondents and non-respondents to the questionnaire invitations at baseline.

DETAILED DESCRIPTION:
Backgrpund:

The interaction between back pain, multimorbidity, and treatment burden can negatively affect patients' participation in treatment pathways and thus their prognosis. However, this has not been sufficiently investigated. A challenge in data collection through, for example, questionnaires is to ensure representative responses from a patient group with expected high treatment burden and lower health literacy. Selective participation can lead to non-response bias and affect conclusions about the impact of multimorbidity on prognoses for individuals with back pain. Therefore, the aim to investigate whether the number of chronic diseases, the treatment burden associated with multimorbidity, and health-related quality of life contribute to non-response bias in this specific population group.

Objectives:

The objectives of this study will be threefold:

1. To examine baseline differences in number of chronic diseases, treatment burden and health-related quality of life among individuals categorized into groups based on their response patterns at baseline.
2. To examine the differences between the aforementioned groups over time (baseline, 3 months, and 6 months).
3. Assess differences in age and sex distribution between responders and non-responders referred for assessment of back pain to questionnaires evaluating their condition.

Through these methods, the aim to uncover any potential non-response bias, which can provide insights for future research. This examination will aid in determining the most effective approach to investigating the influence of multimorbidity on individuals with back pain.

Methods:

In this observational cohort study, data is gathered from patients referred to the Rheumatology Department of Aalborg University Hospital for back pain. Conducted from June 2023 to April 2024, the study recruits participants through electronic links and reminders via E-Boks. Information is sourced from three channels: the department's booking plan (providing details on age and gender of non-responding patients), medical records, and electronic questionnaires. Patient-reported outcomes are collected at baseline, and during 3- and 6-month follow-ups using REDCap.

Patient characteristics include:

* From electronic questionnaire: smoking habits, alcohol consumption, Body mass index, highest achieved education, marital status and work status.
* From medical records: sex, chronic health conditions and use of pain medication,
* Please refer to the section "outcome measures" for details regarding the PROMS.

In this study, multimorbidity is defined as the simultaneous presence of at least two chronic conditions within an individual. The percentage of patients meeting these criteria will be reported, along with a table detailing the frequency of each specific disease.

The patients referred to the department during the time period will be divided into a total of 5 groups.

Group 1) Patients who responded to the first invitation to participate Group 2) Patients who responded to the second invitation to participate Group 3) Patients who responded to the third invitation to participate

In addition, two groups are formed:

Group 4) Patients who dit not respond to any inviations to participate Group 5) an amalgamation of people from the three groups above

Statistical analyses:

Aim 1) To assess baseline differences between groups 1,2 and 3 one-way ANOVA with number of diseases as primary outcome and MTBQ and EQ-5D-5L as secondary outcomes will be employed.

Aim 2) To assess between-group differences at baseline, 3- and 6 months follow up a repeated measurement analysis (RM ANOVA) will be employed with number of diseases as primary outcome and MTBQ and EQ-5D-5L as secondary outcomes.

Additionally, patient characteristics across the three groups will be presented in a table, with appropriate statistical tests used to measure baseline differences (e.g., chi-square test for categorical variables). Results of the repeated measures ANOVA will be visually depicted using bar charts accompanied by error bars.

Imputation will be carried out for missing data if considered appropriate.

Additionally, chi-square test will be employed to assess any differences between group 4 and 5 in terms of gender distrubution. Unpaired t-test will be employed to assess any difference between group 4 and 5 in terms of age.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above
* Diagnosed with neck or back pain and the diagnosis was established by or confirmed by a rheumatologist (clinical expert opinion)
* Speak, read and understand Danish

Exclusion Criteria:

* Withdraw consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals referred for spinal pain to Aalborg University Hospital's Department of Rheumatology between 1st of June 2023 to 1st of March 2024, were invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Multimorbidity Treatment Burden Questionnaire (MTBQ). | This PROM is collected at baseline, 3- and 6 month follow up
  The MTBQ is a 10-item self-report measure designed to assess the burden experienced by individuals with multiple health conditions. The ten items cover various aspects of treatment burden, such as managing one's own health, including self-monitoring and lifestyle changes, dealing with medication-related challenges (e.g., adherence and obtaining prescriptions), coordinating healthcare appointments, and managing dependency on others. Each item was scored on a scale ranging from 0 to 100. A higher total score on the questionnaire indicates a higher burden. The MTBQ has been shown to possess good content validity, construct validity, reliability, and responsiveness and has a valid version in Danish.

SECONDARY OUTCOMES:
Health-related quality of life (EQ-5D-5L) | This PROM is collected at baseline, 3- and 6 months follow up
  A measure of health-related quality of life. The EQ-5D-5L assesses health status across five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension was rated on a five-point ordinal scale ranging from 1 (indicating no problems) to 5 (indicating extreme difficulties). The questionnaire provides a reliable and valid measure of general health and quality of life and is a valid and responsive quality of life scale for patients with chronic low back pain.The minimal important difference for this outcome varies depending on the condition.

OTHER OUTCOMES:
Brief Pain Inventory - Short form | This PROM is collected at baseline, 3- and 6 months follow up
  The Brief Pain Inventory (BPI) is considered the secondary outcome variable. The questionnaire assesses pain in two dimensions: pain intensity and pain interference with function, mood, sleep, and social life, and is a recommended core outcome measure in clinical trials of chronic pain. All items are scored from 0-10, with 0 indicating no pain or interference and 10 indicating worst imaginable pain/completely interference. Hence the sum 0-40 is averaged between the four items about pain intensity, and the sum 0-70 is averaged between the seven items about pain interference.
Insomnia Severity Index | This PROM is collected at baseline, 3- and 6 months follow up
  To assess the patient's sleep quality, the Insomnia Severity Index (ISI) will be utilized. ISI includes seven questions that measure the severity of insomnia experienced over the past two weeks. Respondents assess the severity of difficulties in falling asleep, staying asleep, waking up too early, satisfaction with current sleep, as well as the degree of concern or anxiety caused by sleep problems. Additionally, the impact of sleep difficulties on daytime functioning and whether others notice any impairment related to the sleep issue are also addressed. A 5-point Likert scale (0-4) is used to rate the severity of each area based on the individual's experience. The total score ranges from 0 to 28, where a higher score indicates a greater severity of insomnia.
Patient Health Questionnaire | This PROM is collected at baseline, 3- and 6 months follow up
  The PHQ-2 assesses the frequency of depressed mood and anhedonia over the past two weeks, resulting in a sum score ranging from 0 to 6 points. A score of 3 points indicates a sensitivity of 82.9% and a specificity of 90.0% for major depressive disorder.
Generalized Anxiety Disorder | This PROM is collected at baseline, 3- and 6 months follow up
  Symptoms of anxiety were assessed using the Generalized Anxiety Disorder 2 (GAD-2), which comprises the first two questions of the GAD-7. Patients rated their levels of nervousness, anxiety, or worry, along with their ability to control worrying over the past two weeks. Responses were scored from 0 to 3, resulting in a total score ranging from 0 to 6, with higher scores indicating more pronounced symptoms of anxiety. GAD-2 is considered a covariate.
Work ability score | This PROM is collected at baseline, 3- and 6 months follow up
  The Work Ability Score (WAS) is a single item of the Work Ability Index (WAI), which demonstrates a strong correlation with WAI, revealing similar associations with sick leave, health, and symptoms. In addition, previous research underscores the WAI as a significant prognostic factor for return to work among individuals on long-term sick leave due to pain. In this context, WAS is employed as a predictor for return to work.The scale is scored from 0-10, with higher scores indicating higher self-percieved work ability compared with life time best

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark